CLINICAL TRIAL: NCT00877786
Title: Optimizing Technology in the Treatment of Bulimia Nervosa
Brief Title: Online Cognitive Behavioral Therapy for Bulimia Nervosa
Acronym: CBT4BN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cynthia Bulik, PhD, Distinguished Professor of Eating Disorders, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-2002; R01MH080065-01A1 (NIH)
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Bulimia Nervosa
MeSH Terms: conditions — Bulimia Nervosa | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Face-to-face group therapy (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Group Therapy
- Online chat group therapy (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Group Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Group Therapy — Cognitive behavioral therapy (CBT) is a form of psychotherapy that addresses the links between thoughts, emotions and behaviors.
  Other Names: CBT, Cognitive Behavioral Therapy

SUMMARY:
Cognitive Behavioral Therapy for Bulimia Nervosa (CBT4BN) is a research program funded by the National Institute of Mental Health and conducted by the UNC Eating Disorders Program and the University of Pittsburgh Medical Center. Cognitive Behavioral Therapy (CBT) is an evidence-based treatment and the gold-standard for treating bulimia nervosa. The current study aims to compare two forms of CBT: face-to-face group therapy and online group therapy via cbt4bn.org.

DETAILED DESCRIPTION:
All treatment is conducted by trained professionals from either the UNC Eating Disorders Program (in Chapel Hill) or Western Psychiatric Institute (in Pittsburgh) who are experienced in the treatment of eating disorders.

Participants will participate in 16 1.5 hour long group sessions of group CBT over 20 weeks. Groups will include 5-8 participants, one or two co-therapists, and two sessions by a registered dietitian. Participants will be expected to complete self-monitoring forms which assess their mood and behavior. Groups will either take place face-to-face or online in a therapist-moderated chat group.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for BN
* Internet access at home
* Either off psychotropic medication for at least one month or on a stable dose of psychotropic medication

Exclusion Criteria:

* Any major medical condition that would interfere with treatment or require alternative treatment
* Alcohol or drug dependence in the last three months
* Current significant suicidal ideation
* Developmental disability that would impair the ability to use the internet program effectively
* Psychosis, including schizophrenia, or bipolar I disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2008-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Abstinence from binge/purge episodes | 12 months

SECONDARY OUTCOMES:
Reduction of binge/purge episodes | 12 months
Maintenance of behavior change | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Bulik, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Marsha Marcus, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Watson HJ, McLagan N, Zerwas SC, Crosby RD, Levine MD, Runfola CD, Peat CM, Moessner M, Zimmer B, Hofmeier SM, Hamer RM, Marcus MD, Bulik CM, Crow SJ. Cost-Effectiveness of Internet-Based Cognitive-Behavioral Treatment for Bulimia Nervosa: Results of a Randomized Controlled Trial. J Clin Psychiatry. 2018 Jan/Feb;79(1):16m11314. doi: 10.4088/JCP.16m11314. PMID 29228517
- [Derived] Levinson CA, Zerwas S, Calebs B, Forbush K, Kordy H, Watson H, Hofmeier S, Levine M, Crosby RD, Peat C, Runfola CD, Zimmer B, Moesner M, Marcus MD, Bulik CM. The core symptoms of bulimia nervosa, anxiety, and depression: A network analysis. J Abnorm Psychol. 2017 Apr;126(3):340-354. doi: 10.1037/abn0000254. Epub 2017 Mar 9. PMID 28277735